CLINICAL TRIAL: NCT04174534
Title: DEGENERATIVE DISC DISEASE TREATED BY DECOMPRESSION AND ARTHRODESIS USING A PEEK-TITANIUM POLYAXIAL INTERSPINOUS POSTERIOR FUSION DEVICE: ROMEO®2 PAD. 2 YEARS PROSPECTIVE FOLLOW-UP
Brief Title: ROMEO®2 PAD. 2 YEARS PROSPECTIVE FOLLOW-UP
Acronym: ROMEO 2 PAD FR
Status: Terminated | Type: Observational
Why Stopped: Weak enrollment rate and sanitary situation
Sponsor: Spineart SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P54_CLD004
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed as a post-marketing observational, controlled, prospective, non-inferiority study where the efficacy and safety of the Degenerative Disc Disease treatment by arthrodesis using PEEK(PolyEtherEtherKetone)-Titanium polyaxial interspinous posterior fusion device ROMEO®2 PAD will be compared to the gold standard treatment by instrumented circumferential arthrodesis.

The primary study aim is to evaluate functional improvement at 1 and 2 years after surgery. The fusion at 1 year and 2 years post-surgery, the short and long- term clinical and neurological success and patient related health status satisfaction will also be evaluated.

DETAILED DESCRIPTION:
Lumbar spine fusion is the gold standard technique for the treatment of low-back pain due to various spinal pathologies mostly related to degenerative conditions. Pedicle-screws constructs are widely used to achieve a strong fixation but may be associated with potential complications.

ROMEO® 2 PAD is composed of two polyaxial titanium teethed plates to adapt to anatomical variations, one step locking mechanism and a radiolucent polymer cylinder.

The ROMEO®2 PAD is a posterior non pedicle supplemental fixation device intended for use in combination with an inter-somatic device, to achieve fusion at single or multilevel in the lumbar spine (L1-S1 inclusive). A range of six heights (from 8 to 18mm) are designed to fit anatomical variations. It is intended for plate fixation to the spinous process for the purpose of achieving spinal fixation.

The main objective of the study is the evaluation of functional improvement as measured by changes in Oswestry Disability Index (ODI) at 12 and 24 months after surgery, respectively.

The secondary objectives are:

* Evaluation of fusion rate at 12 and 24 months after surgery, respectively, based on CT scans.
* Evaluation of mobility at the treated level at 12 and 24 months after surgery, respectively, based on ROM (Range of motion) assessed using dynamic lumbar flexion-extension radiography.
* Evaluation of functional capacities post-surgery, as measured by ODI. Comparison between preoperative status and controls at 6 weeks, 6 months after surgery, respectively.
* Evaluation of Health-related Quality of Life (HR-QOL) improvement and patient satisfaction, as measured by SF-36 (Short Form 36) scores, the physical (PCS) and mental (MCS) components; comparison between preoperative status and controls at 6 weeks, 6, at 12 and 24 months after surgery, respectively.
* Evaluation of low back and legs pain as measured by Visual Analogue Scale (VAS) (changes in VAS scores): comparison between preoperative status and controls at 6 weeks, 6, 12 and 24 months after surgery, respectively.

ELIGIBILITY:
Inclusion Criteria:

Surgical treatment of stenosis and Grade I degenerative spondylolisthesis, secondary to lumbar degenerative disc disease at one level between L1 and L5 in skeletally mature patients

Exclusion Criteria:

* Vertebral traumatic lesions including dislocation;
* Insufficient vertebral body bone quality;
* Severe osteoporosis;
* Bone tumor in the region of the implant;
* Spondylolysis;
* Lytic spondylolisthesis;
* Degenerative spondylolisthesis Grade II or more;
* Mental illness or inadequate patient activity;
* Infection;
* Vascular disorders or illness;
* Pregnancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature patients with stenosis and Grade I degenerative spondylolisthesis, secondary to lumbar degenerative disc disease, indicated for treatment with Romeo 2 PAD at one level between L1 and S1.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
ODI | 24 months
  Absolute change in ODI at 12 and 24 months post-operative compared to baseline (pre-operative status)

CONTACTS AND LOCATIONS:
Overall Officials: Dervilla Bermingham, MSc, Study Director — Spineart SA
Locations (3):
- France (3):
  - Hôpital de la Timone, Marseille
  - CHU Gui de Chauliac, Montpellier
  - Clinique St Jean, Montpellier

IPD SHARING:
Plan to Share IPD: No